CLINICAL TRIAL: NCT02901431
Title: A Phase II Multi-Center, Randomized, Double-Blind, 24-Week, Parallel Group, Placebo-Controlled Study to Investigate the Efficacy and Safety of Balovaptan (RO5285119) in Children and Adolescents Age 5-17 With Autism Spectrum Disorder (ASD)
Brief Title: A Study to Investigate the Efficacy and Safety of Balovaptan (RO5285119) in Participants With Autism Spectrum Disorder (ASD)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The 24-week analysis indicated no clinical or statistical benefit for the primary endpoint for the overall study population. No new safety concerns identified.
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BP30153
Record Dates: First submitted 2016-09-12; First posted 2016-09-15 (Estimated); Results first posted 2021-02-08 (Actual); Last update posted 2021-02-08 (Actual); Status verified 2021-01

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Placebo (Placebo Comparator): Participants received a matching placebo orally. Approximate treatment duration was up to 24 weeks.
  Interventions: Drug: Placebo
- Balovaptan (RO5285119) 10 mg/d equivalent (Experimental): Participants received age-adjusted total daily oral dose approximately equivalent to the adult dose of 10 milligrams per day (mg/d) of balovaptan (RO5285119). Approximate treatment duration was up to 24 weeks (up to 52 additional weeks for those enrolled in the OLE).
  Interventions: Drug: RO5285119
- Balovaptan (RO5285119) 4 mg/d equivalent (Experimental): Participants received age-adjusted total daily oral dose approximately equivalent to the adult dose of 4 mg/d of balovaptan (RO5285119). Approximate treatment duration was up to 24 weeks. This arm is open only to those participants enrolled prior to Version 6 of the study protocol.
  Interventions: Drug: RO5285119

INTERVENTIONS:
Drug: Placebo — Participants received a matching placebo orally. Approximate treatment duration was up to 24 weeks.
  Arms: Placebo
Drug: RO5285119 — Participants received age-adjusted total daily oral dose approximately equivalent to the adult doses of either 4 mg/d or 10 mg/d of balovaptan (RO5285119). Approximate treatment duration was up to 24 weeks (up to 52 additional weeks for those enrolled in the OLE).
  Arms: Balovaptan (RO5285119) 10 mg/d equivalent; Balovaptan (RO5285119) 4 mg/d equivalent

SUMMARY:
For participants enrolled prior to Version 6 of the protocol: This was a Phase II multi-center, randomized, double-blind, 24-week, 3-arm, parallel group, placebo-controlled study to investigate the efficacy, safety, and pharmacokinetics of balovaptan in children and adolescents aged 5-17 years with ASD who are high functioning (intelligence quotient [IQ] greater than or equal to [>=] 70).

For participants enrolled according to Version 6 of the protocol: This was a Phase II multi-center, randomized, double-blind, 24-week, parallel group, placebo-controlled, 2-arm study with participants assigned either to a 10 milligram (mg) or equivalent dose of balovaptan, or placebo. All other study parameters remained as stated above.

There are three parts to this study: PK Part (Study part 1) included up to 8 weeks of treatment, Main Treatment Part (Study part 2) included 24 week of treatment, and the Open Label Extension Part (Study part 3) included Week 24 to Week 76 of treatment.

All participants that completed the 24-week treatment period were eligible to participate in an optional 52-week open-label extension (OLE) during which they received balovaptan treatment.

ELIGIBILITY:
Inclusion Criteria:

* Fluent in English
* Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) criteria for ASD or International Statistical Classification of Diseases and Related Health Problems, 10th revision (ICD10) criteria for Autism diagnosis confirmed by Autism Diagnostic Observational Schedule (ADOS-2) criteria
* Social Responsiveness Scale, second edition (SRS-2) (T-score) >= 66
* Clinical Global Impressions of Severity (CGI-S) >= 4 (moderately ill) at screening
* IQ >= 70 as assessed by Wechsler Abbreviated Scale of Intelligence Scale: Second Edition (WASI-II) or Wechsler Preschool and Primary Scale of Intelligence: Fourth Edition (WPPSI-IV) intelligence test
* Language, hearing, and vision compatible with the study measurements as judged by the investigator

Inclusion Criteria for the OLE:

* Have completed the blinded treatment phase of the study OR were required to stop dosing at or before Week 8
* Have no adverse events that would prohibit starting the OLE

Exclusion Criteria:

* Initiation of a major change in psychosocial intervention (including investigational) within 4 weeks prior to screening
* Unstable or uncontrolled clinically significant psychiatric and/or neurological disorder that may interfere with the safety or efficacy endpoints
* Known personal or family history of cerebral aneurysm
* Risk of suicidal behavior
* Seizure within the past 6 months
* Medical history of alcohol or substance abuse/dependence
* Concurrent cardio-vascular disease not considered well controlled by the Investigator
* Clinically significant abnormality on electrocardiogram at screening
* Concomitant disease or condition (pulmonary, gastro-intestinal, hepatic, renal, metabolic, immunological system, or obesity that could interfere with the conduct of the study
* Evidence for current gastro-intestinal bleeding, e.g., active stomach ulcer disease
* History of coagulopathies, bleeding disorders, or blood dyscrasias
* Positive serology for hepatitis B (HBV), hepatitis C (HCV), human immunodeficiency virus (HIV) 1, or HIV 2
* Confirmed clinically significant abnormality in parameters of hematology, clinical chemistry, coagulation, or urinalysis
* Medical history of malignancy if not considered cured
* Participation in an investigational drug study within 90 days or 5 times the half-life of the investigational molecule (whichever is longer) prior to randomization
* Loss of blood over 250 milliliters within three months prior to screening
* Allowed medications have not been stable since 4 weeks before screening, and allowed medications for treatment of epilepsy have not been stable since 3 months before screening
* Use of prohibited medications within 2 weeks prior to screening visit or 5 times the half-life prior to randomization (whichever is longer)

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 339 (Actual)
Dates: Start 2016-11-21 (Actual); Primary Completion 2020-04-15 (Actual); Study Completion 2020-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (45):
- United States (45):
  - Harmonex Neuroscience Research, Dothan, Alabama
  - Southwest Autism Research & Resource Center, Phoenix, Arizona
  - NRC Research Institute, Orange, California
  - PCSD Feighner Research, San Diego, California
  - University of California at San Francisco, San Francisco, California
  - Children's Hospital of Colorado, Aurora, Colorado
  - DBA IMMUNOe Int'l Res Center, Centennial, Colorado
  - Yale University / Yale-New Haven Hospital, New Haven, Connecticut
  - Sarkis Clinical Trials, Gainesville, Florida
  - Segal trials, North Miami, Florida
  - Medical Research Group of Central Florida, Orange City, Florida
  - APG- Advanced Psychiatric Group, Orlando, Florida
  - USF Rothman Center, St. Petersburg, Florida
  - Rush University Medical Center, Chicago, Illinois
  - Capstone Clinical Research, Libertyville, Illinois
  - Kennedy Krieger Institute, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston Childrens Hospital, Boston, Massachusetts
  - Massachusetts General Hospital; Lurie Center for Autism, Lexington, Massachusetts
  - UMASS Medical School, Worcester, Massachusetts
  - University of Minnesota; Clin. Neuro Research Unit, Minneapolis, Minnesota
  - St. Charles Psychiatric Associates, Saint Charles, Missouri
  - Midwest Childrens Health Research Institute, Lincoln, Nebraska
  - Center for Autism and the Developing Brain, New York, New York
  - Nathan S. Kline Institute for Psychiatric Research, Orangeburg, New York
  - University of Rochester, Rochester, New York
  - Richmond Behavioral Associates, Staten Island, New York
  - Albert Einstein College of Medicine, The Bronx, New York
  - DUKE SCHOOL OF MEDICINE;Duke Center for Autism and Brain Development, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - University Hospitals, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Cutting Edge Research Group, Oklahoma City, Oklahoma
  - Suburban Research Associates, Media, Pennsylvania
  - Children's Hospital of Philadelphia;Allergy/Immunology Department, Philadelphia, Pennsylvania
  - UPMC Western Psychiatric Institute and Clinic, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - BioBehavioral Research of Austin, PC, Austin, Texas
  - Relaro Medical Trials, Dallas, Texas
  - Red Oak Psychiatry Associates, PA, Houston, Texas
  - Road Runner Research, San Antonio, Texas
  - Northwest Clinical Research Center, Bellevue, Washington
  - Pacific Institute of Medical Sciences, Bothell, Washington
  - Core Clinical Research, Everett, Washington
  - Seattle Children's Research Institute; Psychiatry and Behavioral Medicine, Seattle, Washington

REFERENCES:
- [Derived] Hollander E, Jacob S, Jou R, McNamara N, Sikich L, Tobe R, Smith J, Sanders K, Squassante L, Murtagh L, Gleissl T, Wandel C, Veenstra-VanderWeele J. Balovaptan vs Placebo for Social Communication in Childhood Autism Spectrum Disorder: A Randomized Clinical Trial. JAMA Psychiatry. 2022 Aug 1;79(8):760-769. doi: 10.1001/jamapsychiatry.2022.1717. PMID 35793101

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 339 participants were enrolled from 44 sites in the United States.
Pre-assignment Details: PK review revealed that age-adjusted doses of 4 and 10 mg in 5-17 year olds were not equivalent to target exposure. For the Main Study Part, data was summarised by exposure ranges (tertiles) based on individual participants PK exposure at Week 12, estimated as the average plasma concentration since treatment start. To allow clear analysis by exposure tertiles, participants with dose adjustment were excluded from analysis by tertiles.
Groups:
- PK Part - Placebo: Participants received a matching placebo orally. Approximate treatment duration was up to 8 weeks.
- PK Part - Balovaptan (RO5285119) 4 mg/d Equivalent: Participants received age-adjusted total daily oral dose approximately equivalent to the adult dose of 4 milligrams per day (mg/d) of balovaptan (RO5285119). Approximate treatment duration was up to 8 weeks.
- PK Part - Balovaptan (RO5285119) 10 mg/d Equivalent: Participants received age-adjusted total daily oral dose approximately equivalent to the adult dose of 10 milligrams per day (mg/d) of balovaptan (RO5285119). Approximate treatment duration was up to 8 weeks.
- Main Study Part - Placebo: Participants received a matching placebo orally. Approximate treatment duration was up to 24 weeks in Main Study Part.
- Main Study Part - Low Exposure Tertile; Main Study Part - Medium Exposure Tertile; Main Study Part - High Exposure Tertile: Participants received age-adjusted total daily oral dose approximately equivalent to the adult dose of 4 or 10 milligrams per day (mg/d) of balovaptan (RO5285119). Approximate treatment duration was up to 24 weeks in Main Study Part.
- Main Study Part - Dose Adjusters: Participants with dose adjustment who were excluded from the analysis by tertiles. Participants received age-adjusted total daily oral dose approximately equivalent to the adult dose of 4 or 10 milligrams per day (mg/d) of balovaptan (RO5285119). Approximate treatment duration was up to 24 weeks in Main Study Part.
- Open Label Extension Part - Placebo; Open Label Extension Part - Low Exposure Tertile; Open Label Extension Part - Medium Exposure Tertile; Open Label Extension Part - High Exposure Tertile: Participants received age-adjusted total daily oral dose approximately equivalent to the adult dose of 10 milligrams per day (mg/d) of balovaptan (RO5285119). Approximate treatment duration was up to 52 weeks in Open Label Extension Part.
- Open Label Extension Part - Dose-Adjusters: Participants with dose adjustment who were excluded from the analysis by tertiles. Participants received age-adjusted total daily oral dose approximately equivalent to the adult dose of 10 milligrams per day (mg/d) of balovaptan (RO5285119). Approximate treatment duration was up to 52 weeks in Open Label Extension Part.
Period: PK Part
Arm/Group | PK Part - Placebo | PK Part - Balovaptan (RO5285119) 4 mg/d Equivalent | PK Part - Balovaptan (RO5285119) 10 mg/d Equivalent | Main Study Part - Placebo | Main Study Part - Low Exposure Tertile | Main Study Part - Medium Exposure Tertile | Main Study Part - High Exposure Tertile | Main Study Part - Dose Adjusters | Open Label Extension Part - Placebo | Open Label Extension Part - Low Exposure Tertile | Open Label Extension Part - Medium Exposure Tertile | Open Label Extension Part - High Exposure Tertile | Open Label Extension Part - Dose-Adjusters
Started | 12 | 11 | 15 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 5 | 5 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 7 | 6 | 9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Pending IMC/SOC Dose Confirmation | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Pending dose confirmation | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — 8 weeks of treatment ran out | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Stopped treatment after 8 weeks | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Stopped on Sponsor instruction pending dose confirmation | 1 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Discontinued per Sponsor | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Main Treatment Part
Arm/Group | PK Part - Placebo | PK Part - Balovaptan (RO5285119) 4 mg/d Equivalent | PK Part - Balovaptan (RO5285119) 10 mg/d Equivalent | Main Study Part - Placebo | Main Study Part - Low Exposure Tertile | Main Study Part - Medium Exposure Tertile | Main Study Part - High Exposure Tertile | Main Study Part - Dose Adjusters | Open Label Extension Part - Placebo | Open Label Extension Part - Low Exposure Tertile | Open Label Extension Part - Medium Exposure Tertile | Open Label Extension Part - High Exposure Tertile | Open Label Extension Part - Dose-Adjusters
Started | 0 | 0 | 0 | 112 | 57 | 66 | 66 | 7 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 86 | 50 | 54 | 55 | 7 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 26 | 7 | 12 | 11 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 3 | 3 | 4 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 3 | 1 | 2 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Caregiver | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 18 | 3 | 5 | 6 | 0 | 0 | 0 | 0 | 0 | 0
Period: Open Label Part
Arm/Group | PK Part - Placebo | PK Part - Balovaptan (RO5285119) 4 mg/d Equivalent | PK Part - Balovaptan (RO5285119) 10 mg/d Equivalent | Main Study Part - Placebo | Main Study Part - Low Exposure Tertile | Main Study Part - Medium Exposure Tertile | Main Study Part - High Exposure Tertile | Main Study Part - Dose Adjusters | Open Label Extension Part - Placebo | Open Label Extension Part - Low Exposure Tertile | Open Label Extension Part - Medium Exposure Tertile | Open Label Extension Part - High Exposure Tertile | Open Label Extension Part - Dose-Adjusters
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 68 | 35 | 40 | 46 | 5
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 20 | 11 | 11 | 7 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 48 | 24 | 29 | 39 | 3
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 4 | 0 | 4 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 1 | 1 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Not completed — Study Terminated By Sponsor | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 35 | 12 | 21 | 31 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 5 | 7 | 3 | 1

BASELINE CHARACTERISTICS:
Population: PK Part & Main Part reported separately. 7 patients ("re-starters") are counted twice. PK review revealed age-adjusted doses of 4 & 10 mg in 5-17 year olds weren't equivalent to target exposure. For Main Study Part, data was summarised by exposure ranges (tertiles) based on individual patients PK exposure at Week 12, estimated as average plasma concentration since treatment start. To allow clear analysis by exposure tertiles, patients with dose adjustment were excluded from analysis by tertiles.
Groups:
- PK Part (Study Part 1) - Placebo: Participants received a matching placebo orally. Approximate treatment duration was up to 8 weeks.
- PK Part (Study Part 1) - Balovaptan (RO5285119) 4 mg/d Equivalent: Participants received age-adjusted total daily oral dose approximately equivalent to the adult dose of 4 milligrams per day (mg/d) of balovaptan (RO5285119). Approximate treatment duration was up to 8 weeks.
- PK Part (Study Part 1) - Balovaptan (RO5285119) 10 mg/d Equivalent: Participants received age-adjusted total daily oral dose approximately equivalent to the adult dose of 10 mg/d of balovaptan (RO5285119). Approximate treatment duration was up to 8 weeks.
- Main Study Part (Study Part 2) - Placebo: Participants in the Main Study Part received a matching placebo orally. Approximate treatment duration was up to 24 weeks.
- Main Study Part (Study Part 2) - Low Exposure Tertile: Participants in the Main Study Part in the Low Exposure Tertile received age-adjusted total daily oral dose approximately equivalent to the adult dose of 4 or 10 milligrams per day (mg/d) of balovaptan (RO5285119). Approximate treatment duration was up to 24 weeks.
- Main Study Part (Study Part 2) - Medium Exposure Tertile: Participants in the Main Study Part in the Medium Exposure Tertile received age-adjusted total daily oral dose approximately equivalent to the adult dose of 4 or 10 milligrams per day (mg/d) of balovaptan (RO5285119). Approximate treatment duration was up to 24 weeks.
- Main Study Part (Study Part 2) - High Exposure Tertile: Participants in the Main Study Part in the High Exposure Tertile received age-adjusted total daily oral dose approximately equivalent to the adult dose of 4 or 10 milligrams per day (mg/d) of balovaptan (RO5285119). Approximate treatment duration was up to 24 weeks.
- Main Study Part (Study Part 2) - Dose-Adjusters: Participants with dose adjustment who were excluded from the analysis by tertiles. Participants received age-adjusted total daily oral dose approximately equivalent to the adult dose of 4 or 10 milligrams per day (mg/d) of balovaptan (RO5285119). Approximate treatment duration was up to 24 weeks in Main Study Part.
- Total: Total of all reporting groups
Arm/Group | PK Part (Study Part 1) - Placebo | PK Part (Study Part 1) - Balovaptan (RO5285119) 4 mg/d Equivalent | PK Part (Study Part 1) - Balovaptan (RO5285119) 10 mg/d Equivalent | Main Study Part (Study Part 2) - Placebo | Main Study Part (Study Part 2) - Low Exposure Tertile | Main Study Part (Study Part 2) - Medium Exposure Tertile | Main Study Part (Study Part 2) - High Exposure Tertile | Main Study Part (Study Part 2) - Dose-Adjusters | Total
Number analyzed (Participants) | 12 | 11 | 15 | 112 | 57 | 66 | 66 | 7 | 346
Age, Continuous [Mean (Standard Deviation); unit: Years] — Participants in the PK part of the study. Population: Participants in the PK part of the study.
  Years
    number analyzed (Participants) | 12 | 11 | 15 | 0 | 0 | 0 | 0 | 0 | 38
    (all) | 8.9 (3.8) | 9.9 (3.3) | 10.4 (3.5) |  |  |  |  |  | 9.8 (3.5)
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: Participants in the Main part of the study.
  Years
    number analyzed (Participants) | 0 | 0 | 0 | 112 | 57 | 66 | 66 | 7 | 308
    (all) |  |  |  | 12.5 (3.0) | 13.3 (2.3) | 12.6 (3.0) | 11.8 (3.3) | 12.6 (2.1) | 12.5 (3.0)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Participants in the PK part of the study.
  Participants
    number analyzed (Participants) | 12 | 11 | 15 | 0 | 0 | 0 | 0 | 0 | 38
    Female | 3 | 1 | 4 | 0 | 0 | 0 | 0 | 0 | 8
    Male | 9 | 10 | 11 | 0 | 0 | 0 | 0 | 0 | 30
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Participants in Main Part of study.
  Participants
    number analyzed (Participants) | 0 | 0 | 0 | 112 | 57 | 66 | 66 | 7 | 308
    Female | 0 | 0 | 0 | 17 | 9 | 8 | 11 | 0 | 45
    Male | 0 | 0 | 0 | 95 | 48 | 58 | 55 | 7 | 263
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Participants in the PK part of the study.
  Participants
    number analyzed (Participants) | 12 | 11 | 15 | 0 | 0 | 0 | 0 | 0 | 38
    Hispanic or Latino | 2 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 6
    Not Hispanic or Latino | 10 | 10 | 11 | 0 | 0 | 0 | 0 | 0 | 31
    Unknown or Not Reported | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Participants in the main part of the study.
  Participants
    number analyzed (Participants) | 0 | 0 | 0 | 112 | 57 | 66 | 66 | 7 | 308
    Hispanic or Latino | 0 | 0 | 0 | 17 | 7 | 8 | 6 | 0 | 38
    Not Hispanic or Latino | 0 | 0 | 0 | 93 | 49 | 58 | 59 | 7 | 266
    Unknown or Not Reported | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Participants in PK part of the study.
  Participants
    number analyzed (Participants) | 12 | 11 | 15 | 0 | 0 | 0 | 0 | 0 | 38
    American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Asian | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Black or African American | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 3
    White | 11 | 9 | 10 | 0 | 0 | 0 | 0 | 0 | 30
    More than one race | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
    Unknown or Not Reported | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants] — Participants in Main Part of study Population: Participants in Main Part of study.
  Participants
    number analyzed (Participants) | 0 | 0 | 0 | 112 | 57 | 66 | 66 | 7 | 308
    American Indian or Alaska Native | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
    Asian | 0 | 0 | 0 | 5 | 3 | 7 | 3 | 0 | 18
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
    Black or African American | 0 | 0 | 0 | 4 | 1 | 4 | 5 | 0 | 14
    White | 0 | 0 | 0 | 93 | 46 | 54 | 51 | 6 | 250
    More than one race | 0 | 0 | 0 | 9 | 5 | 1 | 5 | 1 | 21
    Unknown or Not Reported | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Vineland™-II Adaptive Behavior Scale Two Domain Composite (2DC) Score at Week 24 for Balovaptan (R05285119) 10 mg Equivalent Compared to Placebo
Description: Vineland™-II Adaptive Behavior Scales 2-Domain Composite (2DC) Score is defined as mean of the Communication domain standard score & Socialization domain standard score. If any of the 2 individual domain standard scores is missing 2DC score is not computed. Vineland™-II is an instrument that measures communication, daily living skills, socialization, motor skills and maladaptive behavior of individuals with developmental disabilities. Survey Interview Form will be administered to a subject's reliable caregiver in this study, during which the rater or clinician will ask to the caregiver open ended questions relating to the subject's activities and behavior. Standardized scores on the Adaptive behavior composite range from 20-160 with higher scores indicating better functioning. Mixed model with repeated measures (MMRM) was used for analysis with assessments at baseline, week 12 and week 24.
Time Frame: Baseline, Week 24
Population: Efficacy Inferential Population included participants that were divided by randomized treatment and included participants taking balovaptan 10 mg equivalent dose and participants from the concurrently randomized placebo group in the corresponding randomization stage. Participants with dose adjustments or interruptions, or who were on a different dose than the final dose for their age group, were excluded.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Groups:
- Balovaptan (RO5285119) 10 mg/d Equivalent: Participants received age-adjusted total daily oral dose approximately equivalent to the adult dose of 10 milligrams per day (mg/d) of balovaptan (RO5285119). Approximate treatment duration was up to 24 weeks.
Arm/Group | Placebo | Balovaptan (RO5285119) 10 mg/d Equivalent
Number analyzed (Participants) | 81 | 86
Score on a scale | 2.34 (1.15) | 2.17 (1.11)
Statistical Analysis 1: Comparison: Placebo vs Balovaptan (RO5285119) 10 mg/d Equivalent; Test type: Superiority; p = 0.911, Mixed Models Analysis; Difference in Adjusted LSMeans = -0.16, 90% CI 2-sided [-2.56 to 2.23]

2. Secondary Outcome: Change From Baseline in Vineland™-II Composite Standard Score After 12 Weeks and 24 Weeks of Treatment for Balovaptan (R05285119) 10 mg Equivalent Compared to Placebo
Description: The Vineland™-II is an instrument that measures communication, daily living skills, socialization, motor skills (only in children up to 6 years) and maladaptive (not assessed in this study) behavior of individuals with developmental disabilities. The Survey Interview Form (i.e., semi -structured interview) will be administered to a subject's reliable caregiver in this study, during which the rater or clinician will ask to the caregiver open ended questions relating to the subject's activities and behavior. Domain scores will be obtained for the individual domains of Socialization, Communication, Daily Living Skills, and motor skills (up to 6 years only) and used to calculate the Vineland-II Adaptive Behavior Composite score. Standardized scores on the Adaptive behavior composite range from 20-160 with higher scores indicating better functioning.
Time Frame: Baseline, Weeks 12 and 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | Balovaptan (RO5285119) 10 mg/d Equivalent
Number analyzed (Participants) | 81 | 86
Score on a scale
  Week 12 | 1.45 (1.07) | 1.74 (1.04)
  Week 24 | 2.20 (1.19) | 1.97 (1.15)
Statistical Analysis 1: Comparison: Placebo vs Balovaptan (RO5285119) 10 mg/d Equivalent; Week 12; Test type: Superiority; Difference in adjused LSMean = 0.29, 90% CI 2-sided [-1.85 to 2.43]
Statistical Analysis 2: Comparison: Placebo vs Balovaptan (RO5285119) 10 mg/d Equivalent; Week 24; Test type: Superiority; Difference in adjusted LSMean = -0.23, 90% CI 2-sided [-2.67 to 2.22]

3. Secondary Outcome: Change From Baseline in Vineland™-II Adaptive Behavior Scale Communication, Socialization, and Daily Living Skills Domain Standard Scores at Weeks 12 and 24 for Balovaptan (R05285119) 10 mg Equivalent Compared to Placebo
Description: The Vineland™-II is an instrument that measures communication, daily living skills, socialization, motor skills (only in children up to 6 years) and maladaptive (not assessed in this study) behavior of individuals with developmental disabilities. The Survey Interview Form (i.e., semi -structured interview) will be administered to a subject's reliable caregiver in this study, during which the rater or clinician will ask to the caregiver open ended questions relating to the subject's activities and behavior. Domain scores will be obtained for the individual domains of Socialization, Communication, and Daily Living Skills. Standardized scores on the domains range from 20-160 with higher scores indicating better functioning. Measure Type is Adjusted least-squares means.
Time Frame: Baseline, Weeks 12 and 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | Balovaptan (RO5285119) 10 mg/d Equivalent
Number analyzed (Participants) | 81 | 86
Score on a scale
  Communication Domain Standard Score, Week 12 | 1.86 (1.06) | 1.64 (1.03)
  Communication Domain Standard Score, Week 24 | 1.51 (1.13) | 2.21 (1.09)
  Socialization Domain Standard Score, Week 12 | 1.69 (1.31) | 2.20 (1.26)
  Socialization Domain Standard Score, Week 24 | 2.87 (1.50) | 2.26 (1.45)
  Daily Living Skills Domain Standard Score, Week 12 | -0.01 (1.38) | 2.13 (1.35)
  Daily Living Skills Domain Standard Score, Week 24 | 1.44 (1.49) | 1.61 (1.45)
Statistical Analysis 1: Comparison: Placebo vs Balovaptan (RO5285119) 10 mg/d Equivalent; Communication Domain Standard Score, Week 12; Test type: Superiority; Difference in adjusted LSMean = -0.22, 90% CI 2-sided [-2.36 to 1.92]
Statistical Analysis 2: Comparison: Placebo vs Balovaptan (RO5285119) 10 mg/d Equivalent; Communication Domain Standard Score, Week 24; Test type: Superiority; Difference in adjusted LSMean = 0.71, 90% CI 2-sided [-1.60 to 3.02]
Statistical Analysis 3: Comparison: Placebo vs Balovaptan (RO5285119) 10 mg/d Equivalent; Socialization Domain Standard Score, Week 12; Test type: Superiority; Difference in adjusted LSMean = 0.51, 90% CI 2-sided [-2.10 to 3.12]
Statistical Analysis 4: Comparison: Placebo vs Balovaptan (RO5285119) 10 mg/d Equivalent; Test type: Superiority — Socialization Domain Standard Score, Week 24; Difference in adjusted LSMean = -0.61, 90% CI 2-sided [-3.74 to 2.51]
Statistical Analysis 5: Comparison: Placebo vs Balovaptan (RO5285119) 10 mg/d Equivalent; Test type: Superiority — Daily Living Skills Domain Standard Score, Week 12; Difference in adjusted LSMean = 2.14, 90% CI 2-sided [-0.63 to 4.90]
Statistical Analysis 6: Comparison: Placebo vs Balovaptan (RO5285119) 10 mg/d Equivalent; Test type: Superiority — Daily Living Skills Domain Standard Score, Week 24; Differences in adjusted LSMean = 0.18, 90% CI 2-sided [-2.87 to 3.22]

4. Secondary Outcome: Proportion of Subjects With >=6 Points Improvement in the Vineland-II 2DC Score for Balovaptan (R05285119) 10 mg Equivalent Compared to Placebo
Description: Vineland™-II Adaptive Behavior Scales 2-Domain Composite (2DC) Score is defined as mean of the Communication domain standard score & Socialization domain standard score. If any of the 2 individual domain standard scores is missing 2DC score is not computed. Vineland™-II is an instrument that measures communication, daily living skills, socialization, motor skills and maladaptive behavior of individuals with developmental disabilities. Survey Interview Form will be administered to a subject's reliable caregiver in this study, during which the rater or clinician will ask to the caregiver open ended questions relating to the subject's activities and behavior. Domain scores will be obtained for the individual domains of Socialization, Communication, Daily Living Skills, and motor skills and used to calculate the Vineland™-II Adaptive Behavior Composite score. Standardized scores on the Adaptive behavior composite range from 20-160 with higher scores indicating better functioning.
Time Frame: Baseline, Weeks 12 and 24
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Balovaptan (RO5285119) 10 mg/d Equivalent
Number analyzed (Participants) | 66 | 70
Percentage of participants
  Week 12 | 30.3 | 27.1
  Week 24: number analyzed (Participants) | 61 | 67
  Week 24 | 34.4 | 32.8

5. Secondary Outcome: Change From Baseline in Clinical Global Impressions-Severity (CGI-S) Score at Weeks 12 and 24 for Balovaptan (R05285119) 10 mg Equivalent Compared to Placebo
Description: The CGI-S reflects the rater's impression of the subject's current autism severity on a 7-point scale ranging from no symptoms (1) to very severe symptoms (7). Changes in CGI-S score were calculated as increase or decrease in absolute CGI-S scores between Baseline and Weeks 12 and 24.
Time Frame: Baseline, Weeks 12 and 24
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Balovaptan (RO5285119) 10 mg/d Equivalent
Number analyzed (Participants) | 67 | 74
Percentage of participants
  -3 (Very much improved), Week 12 | 1.5 | 0
  -2 (Much improved), Week 12 | 1.5 | 2.7
  -1 (Minimally improved), Week 12 | 31.3 | 31.1
  0 (No change), Week 12 | 65.7 | 63.5
  +1 (Minimally worse), Week 12 | 0 | 2.7
  +2 (Much worse), Week 12 | 0 | 0
  +3 (Very Much worse), Week 12 | 0 | 0
  -3 (Very much improved), Week 24: number analyzed (Participants) | 62 | 69
  -3 (Very much improved), Week 24 | 1.6 | 0
  -2 (Much improved), Week 24: number analyzed (Participants) | 62 | 69
  -2 (Much improved), Week 24 | 6.5 | 4.3
  -1 (Minimally improved), Week 24: number analyzed (Participants) | 62 | 69
  -1 (Minimally improved), Week 24 | 32.3 | 31.9
  0 (No change), Week 24: number analyzed (Participants) | 62 | 69
  0 (No change), Week 24 | 59.7 | 63.8
  +1 (Minimally worse), Week 24: number analyzed (Participants) | 62 | 69
  +1 (Minimally worse), Week 24 | 0 | 0
  +2 (Much worse), Week 24: number analyzed (Participants) | 62 | 69
  +2 (Much worse), Week 24 | 0 | 0
  +3 (Very much worse), Week 24: number analyzed (Participants) | 62 | 69
  +3 (Very much worse), Week 24 | 0 | 0

6. Secondary Outcome: Change From Baseline in Ohio Autism Clinical Impressions Scale-Severity (OACIS-S) Score at Weeks 12 and 24 for Balovaptan (R05285119) 10 mg Equivalent Compared to Placebo
Description: The OACIS-S is a 10-item, clinician-completed measures based upon interview and/or observation. The OACIS-S assess severity and improvement, respectively, in social interaction, aberrant behavior, repetitive or ritualistic behavior, verbal communication, nonverbal communication skills, hyperactivity and inattention, anxiety and fearfulness, sensory sensitivities, restricted and narrow interests, and a global rating of autism. Each item of the OACIS-S is rated on a 7-point scale ranging from no symptoms (1) to very severe symptoms (7). Changes in CGI-S score were calculated as increase or decrease in absolute CGI-S scores between Baseline and Weeks 12 and 24.
Time Frame: Baseline, Weeks 12 and 24
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Balovaptan (RO5285119) 10 mg/d Equivalent
Number analyzed (Participants) | 67 | 73
Percentage of participants
  -3 (Very much improved), Week 12 | 3.0 | 0
  -2 (Much improved), Week 12 | 6.0 | 6.8
  -1 (Minimally improved), Week 12 | 28.4 | 34.2
  0 (No change), Week 12 | 59.7 | 57.5
  +1 (Minimally worse), Week 12 | 3.0 | 1.4
  +2 (Much worse), Week 12 | 0 | 0
  +3 (Very much worse), Week 12 | 0 | 0
  -3 (Very much improved), Week 24: number analyzed (Participants) | 62 | 67
  -3 (Very much improved), Week 24 | 6.5 | 0
  -2 (Much improved), Week 24: number analyzed (Participants) | 62 | 67
  -2 (Much improved), Week 24 | 8.1 | 7.5
  -1 (Minimally improved), Week 24: number analyzed (Participants) | 62 | 67
  -1 (Minimally improved), Week 24 | 33.9 | 28.4
  0 (No change), Week 24: number analyzed (Participants) | 62 | 67
  0 (No change), Week 24 | 48.4 | 61.2
  +1 (Minimally worse), Week 24: number analyzed (Participants) | 62 | 67
  +1 (Minimally worse), Week 24 | 3.2 | 3.0
  +2 (Much worse), Week 24: number analyzed (Participants) | 62 | 67
  +2 (Much worse), Week 24 | 0 | 0
  +3 (Very much worse), Week 24: number analyzed (Participants) | 62 | 67
  +3 (Very much worse), Week 24 | 0 | 0

7. Secondary Outcome: Clinical Global Impressions- Improvement (CGI-I) Score at Weeks 12 and 24 for Balovaptan (R05285119) 10 mg Equivalent Compared to Placebo
Description: The CGI rating scales are tools used to evaluate both the severity of illness and change from baseline. The CGI-I is used to assess the clinical change as compared to symptoms at baseline using a 7-point scale, ranging from very much improved (1) to very much worse (7). For this study modified versions will be used.
Time Frame: Weeks 12 and 24
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Balovaptan (RO5285119) 10 mg/d Equivalent
Number analyzed (Participants) | 67 | 74
Percentage of participants
  1 - Very much improved, Week 12 | 0 | 0
  2 - Much improved, Week 12 | 22.4 | 21.6
  3 - Minimally improved, Week 12 | 49.3 | 35.1
  4 - No change, Week 12 | 22.4 | 43.2
  5 - Minimally worse, Week 12 | 6.0 | 0
  6 - Much worse, Week 12 | 0 | 0
  7 - Very much worse, Week 12 | 0 | 0
  1 - Very much improved, Week 24: number analyzed (Participants) | 62 | 68
  1 - Very much improved, Week 24 | 0 | 4.4
  2 - Much improved, Week 24: number analyzed (Participants) | 62 | 68
  2 - Much improved, Week 24 | 30.6 | 26.5
  3 - Minimally improved, Week 24: number analyzed (Participants) | 62 | 68
  3 - Minimally improved, Week 24 | 48.4 | 30.9
  4 - No change, Week 24: number analyzed (Participants) | 62 | 68
  4 - No change, Week 24 | 19.4 | 36.8
  5 - Minimally worse, Week 24: number analyzed (Participants) | 62 | 68
  5 - Minimally worse, Week 24 | 1.6 | 1.5
  6 - Much worse, Week 24: number analyzed (Participants) | 62 | 68
  6 - Much worse, Week 24 | 0 | 0
  7 - Very much worse, Week 24: number analyzed (Participants) | 62 | 68
  7 - Very much worse, Week 24 | 0 | 0

8. Secondary Outcome: Ohio Autism Clinical Impressions Scale- Improvement (OACIS-I) Score at Weeks 12 and 24 for Balovaptan (R05285119) 10 mg Equivalent Compared to Placebo
Description: The OACIS-I is a 10-item, clinician-completed measures based upon interview and/or observation. The OACIS-I assess severity and improvement, respectively, in social interaction, aberrant behavior, repetitive or ritualistic behavior, verbal communication, nonverbal communication skills, hyperactivity and inattention, anxiety and fearfulness, sensory sensitivities, restricted and narrow interests, and a global rating of autism. The OACIS-I is used to assess the clinical change as compared to symptoms at baseline using a 7-point scale, ranging from very much improved (1) to very much worse (7).
Time Frame: Weeks 12 and 24
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Balovaptan (RO5285119) 10 mg/d Equivalent
Number analyzed (Participants) | 67 | 74
Percentage of participants
  1 - Very much improved, Week 12 | 1.5 | 0
  2 - Much improved, Week 12 | 16.4 | 20.3
  3 - Minimally improved, Week 12 | 38.8 | 25.7
  4 - No change, Week 12 | 40.3 | 54.1
  5 - Minimally worse, Week 12 | 3.0 | 0
  6 - Much worse, Week 12 | 0 | 0
  7 - Very much worse, Week 12 | 0 | 0
  1 - Very much improved, Week 24: number analyzed (Participants) | 62 | 68
  1 - Very much improved, Week 24 | 0 | 2.9
  2 - Much improved, Week 24: number analyzed (Participants) | 62 | 68
  2 - Much improved, Week 24 | 25.8 | 22.1
  3 - Minimally improved, Week 24: number analyzed (Participants) | 62 | 68
  3 - Minimally improved, Week 24 | 46.8 | 25.0
  4 - No change, Week 24: number analyzed (Participants) | 62 | 68
  4 - No change, Week 24 | 25.8 | 50.0
  5 - Minimally worse, Week 24: number analyzed (Participants) | 62 | 68
  5 - Minimally worse, Week 24 | 1.6 | 0
  6 - Much worse, Week 24: number analyzed (Participants) | 62 | 68
  6 - Much worse, Week 24 | 0 | 0
  7 - Very much worse, Week 24: number analyzed (Participants) | 62 | 68
  7 - Very much worse, Week 24 | 0 | 0

9. Secondary Outcome: Change From Baseline in Patient-Reported Pediatric Quality of Life (PedsQL) v4.0 Generic Core Scale After 12 Weeks and 24 Weeks of Treatment for Balovaptan (R05285119) 10 mg Equivalent Compared to Placebo
Description: The Pediatric Quality of Life Inventory PedsQL™4.0 Generic Core Scale assessment consists of a 23 item questionnaire encompassing 4 core scale domains: Physical Functioning (8 items); Emotional Functioning (5 items); Social Functioning (5 items); and School Functioning (5 items). For children aged 8 years and above, the PedsQL items are scored on a 5 point Likert-type response scale (0=never a problem; 1=almost never a problem; 2=sometimes a problem; 3=often a problem; and 4=almost always a problem). For children aged 5-7 years, scoring is based on a three-point scale (0=Not at all, 2=Sometimes, 4=A lot). Once scored, items will be reverse scored and linearly transformed to a 0-100 scale (0=100, 1=75, 2=50, 3=25, 4=0), so that higher scores indicate better health-related quality of life.
Time Frame: Baseline, Weeks 12 and 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Score on scale
Arm/Group | Placebo | Balovaptan (RO5285119) 10 mg/d Equivalent
Number analyzed (Participants) | 62 | 72
Score on scale
  Change from Baseline at Week 12 | 2.42 (1.49) | 6.16 (1.41)
  Change from Baseline at Week 24: number analyzed (Participants) | 59 | 65
  Change from Baseline at Week 24 | 3.70 (1.50) | 5.98 (1.44)
Statistical Analysis 1: Comparison: Placebo vs Balovaptan (RO5285119) 10 mg/d Equivalent; Week 12; Test type: Superiority; Mixed Models Analysis; Difference of Adjusted LS Means = 3.74, 90% CI 2-sided [0.78 to 6.70]
Statistical Analysis 2: Comparison: Placebo vs Balovaptan (RO5285119) 10 mg/d Equivalent; Week 24; Test type: Superiority; Difference of Adjusted LS means = 2.28, 90% CI 2-sided [-0.73 to 5.29]

10. Secondary Outcome: Change From Baseline in Vineland-II Composite Standard Score in Adolescents and Children Independently at Weeks 12 and 24 for Balovaptan (R05285119) 10 mg Equivalent Compared to Placebo
Description: The Vineland-II is an instrument that measures communication, daily living skills, socialization, motor skills (only in children up to 6 years) and maladaptive (not assessed in this study) behavior of individuals with developmental disabilities. The Survey Interview Form (i.e., semi -structured interview) will be administered to a subject's reliable caregiver in this study, during which the rater or clinician will ask to the caregiver open ended questions relating to the subject's activities and behavior. Domain scores will be obtained for the individual domains of Socialization, Communication, Daily Living Skills, and motor skills (up to 6 years only) and used to calculate the Vineland-II Adaptive Behavior Composite score. Standardized scores on the Adaptive behavior composite range from 20-160 with higher scores indicating better functioning.
Time Frame: Baseline, Weeks 12 and 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Placebo | Balovaptan (RO5285119) 10 mg/d Equivalent
Number analyzed (Participants) | 44 | 48
Score on scale
  5-12 Years Age Group, Absolute Value at Baseline | 73.9 (9.7) | 77.3 (10.9)
  5-12 Years Age Group, Change From Baseline at Week 12: number analyzed (Participants) | 37 | 38
  5-12 Years Age Group, Change From Baseline at Week 12 | 3.6 (8.4) | 1.2 (7.8)
  5-12 Years Age Group, Change From Baseline at Week 24: number analyzed (Participants) | 34 | 37
  5-12 Years Age Group, Change From Baseline at Week 24 | 4.8 (9.1) | 1.0 (8.4)
  13-17 Years Age Group, Absolute Baseline Value: number analyzed (Participants) | 35 | 36
  13-17 Years Age Group, Absolute Baseline Value | 71.0 (10.3) | 73.5 (8.9)
  13-17 Years Age Group, Change From Baseline at Week 12: number analyzed (Participants) | 29 | 32
  13-17 Years Age Group, Change From Baseline at Week 12 | 1.8 (4.8) | 3.7 (9.4)
  13-17 Years Age Group, Change From Baseline at Week 24: number analyzed (Participants) | 27 | 30
  13-17 Years Age Group, Change From Baseline at Week 24 | 2.7 (8.6) | 3.3 (8.7)

11. Secondary Outcome: Change From Baseline in Vineland-II Adaptive Behavior Scale 2DC Score at Week 12 for Balovaptan (R05285119) 10 mg Equivalent Compared to Placebo
Description: The Vineland-II is an instrument that measures communication, daily living skills, socialization, motor skills (only in children up to 6 years) and maladaptive (not assessed in this study) behavior of individuals with developmental disabilities. The Survey Interview Form (i.e., semi -structured interview) will be administered to a subject's reliable caregiver in this study, during which the rater or clinician will ask to the caregiver open ended questions relating to the subject's activities and behavior. Domain scores will be obtained for the individual domains of Socialization, Communication, Daily Living Skills, and motor skills (up to 6 years only) and used to calculate the Vineland-II Adaptive Behavior Composite score. Standardized scores on the Adaptive behavior composite range from 20-160 with higher scores indicating better functioning. Mixed model with repeated measures (MMRM) was used for analysis.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Score on scale
Arm/Group | Placebo | Balovaptan (RO5285119) 10 mg/d Equivalent
Number analyzed (Participants) | 81 | 86
Score on scale | 1.87 (1.00) | 1.88 (0.97)
Statistical Analysis 1: Comparison: Placebo vs Balovaptan (RO5285119) 10 mg/d Equivalent; Test type: Superiority; p = 0.992, Mixed Models Analysis; Difference in Adjusted LS Means = 0.01, 90% CI 2-sided [-1.99 to 2.01]

12. Secondary Outcome: Percentage of Participants With Adverse Events for Treatment With Balovaptan
Description: PK review revealed that age-adjusted doses of 4 and 10 mg in 5-17 year olds were not equivalent to target exposure. For the Main Study Part, data was summarised by exposure ranges (tertiles) based on individual participants PK exposure at Week 12, estimated as the average plasma concentration since treatment start. To allow clear analysis by exposure tertiles, participants with dose adjustment were excluded from analysis by tertiles.
Time Frame: Baseline to Week 24 and up to Week 76
Population: Safety Population consisted of all participants who received a least one dose of study medication; Used for safety analyses and divided by exposure tertiles.
Measure: Number; unit: Percentage of Participants
Groups:
- Main Study Part, Low Exposure Tertile: Participants in the Main Study Part in the Low Exposure Tertile received age-adjusted total daily oral dose approximately equivalent to the adult dose of 4 or 10 milligrams per day (mg/d) of balovaptan (RO5285119). Approximate treatment duration was up to 24 weeks.
- Main Study Part, Medium Exposure Tertile: Participants in the Main Study Part in the Medium Exposure Tertile received age-adjusted total daily oral dose approximately equivalent to the adult dose of 4 or 10 milligrams per day (mg/d) of balovaptan (RO5285119). Approximate treatment duration was up to 24 weeks.
- Main Study Part, High Exposure Tertile: Participants in the Main Study Part in the High Exposure Tertile received age-adjusted total daily oral dose approximately equivalent to the adult dose of 4 or 10 milligrams per day (mg/d) of balovaptan (RO5285119). Approximate treatment duration was up to 24 weeks.
- Main Study Part (Study Part 2) - All Treated: All participants in the Main Study Part received age-adjusted total daily oral dose approximately equivalent to the adult dose of 4 or 10 milligrams per day (mg/d) of balovaptan (RO5285119). This group includes participants from the low, medium, and high exposure tertiles, as well as the Dose-Adjusters. Approximate treatment duration was up to 24 weeks.
- Open Label Extension Part, Low Exposure Tertile: Participants in the Open Label Extension Part of the study in the Low Exposure Tertile received age-adjusted total daily oral dose approximately equivalent to the adult dose of 10 milligrams per day (mg/d) of balovaptan (RO5285119). Approximate treatment duration was up to 52 weeks.
- Open Label Extension Part, Medium Exposure Tertile: Participants in the Open Label Extension Part of the study in the Medium Exposure Tertile received age-adjusted total daily oral dose approximately equivalent to the adult dose of 10 milligrams per day (mg/d) of balovaptan (RO5285119). Approximate treatment duration was up to 52 weeks in Open Label Extension Part.
- Open Label Extension Part, High Exposure Tertile: Participants in the Open Label Extension Part of the study in the High Exposure Tertile received age-adjusted total daily oral dose approximately equivalent to the adult dose of 10 milligrams per day (mg/d) of balovaptan (RO5285119). Approximate treatment duration was up 52 weeks.
- Open Label Extension Part, All Treated: All participants in the Open Label Extension Part of the study received age-adjusted total daily oral dose approximately equivalent to the adult dose of 10 milligrams per day (mg/d) of balovaptan (RO5285119). This group includes participants from the low, medium, and high exposure tertiles, as well as the Dose-Adjusters. Approximate treatment duration was up to 52 weeks.
Arm/Group | Main Study Part, Low Exposure Tertile | Main Study Part, Medium Exposure Tertile | Main Study Part, High Exposure Tertile | Main Study Part (Study Part 2) - All Treated | Open Label Extension Part, Low Exposure Tertile | Open Label Extension Part, Medium Exposure Tertile | Open Label Extension Part, High Exposure Tertile | Open Label Extension Part, All Treated
Number analyzed (Participants) | 57 | 66 | 66 | 196 | 35 | 40 | 46 | 126
Percentage of Participants | 77.2 | 71.2 | 66.7 | 71.4 | 68.6 | 70.0 | 78.3 | 72.2

ADVERSE EVENTS:
Time Frame: From the first study drug to the data cutoff date: 30 June 2020 (up to 43 months)
Description: PK review revealed that age-adjusted doses of 4 and 10 mg in 5-17 year olds were not equivalent to target exposure. For the Main Study Part, data was summarised by exposure ranges (tertiles) based on individual participants PK exposure at Week 12, estimated as the average plasma concentration since treatment start. To allow clear analysis by exposure tertiles, participants with dose adjustment were excluded from analysis by tertiles.
Groups:
- PK Part (Study Part 1) - Placebo: Participants in the PK Part of the study who received a matching placebo orally. Approximate treatment duration was up to 8 weeks.
- PK Part (Study Part 1) - Balovaptan (RO5285119) 4 mg/d Equivalent: Participants in the PK Part of the study who received age-adjusted total daily oral dose approximately equivalent to the adult dose of 4 milligrams per day (mg/d) of balovaptan (RO5285119). Approximate treatment duration was up to 8 weeks.
- PK Part (Study Part 1) - Balovaptan (RO5285119) 10 mg/d Equivalent: Participants in the PK Part of the study who received age-adjusted total daily oral dose approximately equivalent to the adult dose of 10 milligrams per day (mg/d) of balovaptan (RO5285119). Approximate treatment duration was up to 8 weeks.
- Open Label Extension Part (Study Part 3) - Placebo; Open Label Extension Part (Study Part 3) - Low Exposure Tertile; Open Label Extension Part (Study Part 3) - Medium Exposure Tertile; Open Label Extension Part (Study Part 3) - High Exposure Tertile: Participants received age-adjusted total daily oral dose approximately equivalent to the adult dose of 10 milligrams per day (mg/d) of balovaptan (RO5285119). Approximate treatment duration was up to 52 weeks in Open Label Extension Part.
- Open Label Extension Part (Study Part 3) - Dose-Adjusters: Participants with dose adjustment who were excluded from the analysis by tertiles. Participants received age-adjusted total daily oral dose approximately equivalent to the adult dose of 10 milligrams per day (mg/d) of balovaptan (RO5285119). Approximate treatment duration was up to 52 weeks in Open Label Extension Part.
Arm/Group | PK Part (Study Part 1) - Placebo | PK Part (Study Part 1) - Balovaptan (RO5285119) 4 mg/d Equivalent | PK Part (Study Part 1) - Balovaptan (RO5285119) 10 mg/d Equivalent | Main Study Part (Study Part 2) - Placebo | Main Study Part (Study Part 2) - Low Exposure Tertile | Main Study Part (Study Part 2) - Medium Exposure Tertile | Main Study Part (Study Part 2) - High Exposure Tertile | Main Study Part (Study Part 2) - Dose-Adjusters | Open Label Extension Part (Study Part 3) - Placebo | Open Label Extension Part (Study Part 3) - Low Exposure Tertile | Open Label Extension Part (Study Part 3) - Medium Exposure Tertile | Open Label Extension Part (Study Part 3) - High Exposure Tertile | Open Label Extension Part (Study Part 3) - Dose-Adjusters
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/11 | 0/15 | 0/112 | 0/57 | 0/66 | 0/66 | 0/7 | 0/68 | 0/35 | 0/40 | 0/46 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/12 | 1/11 | 0/15 | 4/112 | 1/57 | 0/66 | 1/66 | 0/7 | 2/68 | 0/35 | 0/40 | 2/46 | 0/5
Other Adverse Events (participants affected / at risk) | 7/12 | 7/11 | 7/15 | 58/112 | 34/57 | 31/66 | 34/66 | 5/7 | 35/68 | 21/35 | 25/40 | 27/46 | 3/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PK Part (Study Part 1) - Placebo (N=12) | PK Part (Study Part 1) - Balovaptan (RO5285119) 4 mg/d Equivalent (N=11) | PK Part (Study Part 1) - Balovaptan (RO5285119) 10 mg/d Equivalent (N=15) | Main Study Part (Study Part 2) - Placebo (N=112) | Main Study Part (Study Part 2) - Low Exposure Tertile (N=57) | Main Study Part (Study Part 2) - Medium Exposure Tertile (N=66) | Main Study Part (Study Part 2) - High Exposure Tertile (N=66) | Main Study Part (Study Part 2) - Dose-Adjusters (N=7) | Open Label Extension Part (Study Part 3) - Placebo (N=68) | Open Label Extension Part (Study Part 3) - Low Exposure Tertile (N=35) | Open Label Extension Part (Study Part 3) - Medium Exposure Tertile (N=40) | Open Label Extension Part (Study Part 3) - High Exposure Tertile (N=46) | Open Label Extension Part (Study Part 3) - Dose-Adjusters (N=5)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aggression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intentional self-injury (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PK Part (Study Part 1) - Placebo (N=12) | PK Part (Study Part 1) - Balovaptan (RO5285119) 4 mg/d Equivalent (N=11) | PK Part (Study Part 1) - Balovaptan (RO5285119) 10 mg/d Equivalent (N=15) | Main Study Part (Study Part 2) - Placebo (N=112) | Main Study Part (Study Part 2) - Low Exposure Tertile (N=57) | Main Study Part (Study Part 2) - Medium Exposure Tertile (N=66) | Main Study Part (Study Part 2) - High Exposure Tertile (N=66) | Main Study Part (Study Part 2) - Dose-Adjusters (N=7) | Open Label Extension Part (Study Part 3) - Placebo (N=68) | Open Label Extension Part (Study Part 3) - Low Exposure Tertile (N=35) | Open Label Extension Part (Study Part 3) - Medium Exposure Tertile (N=40) | Open Label Extension Part (Study Part 3) - High Exposure Tertile (N=46) | Open Label Extension Part (Study Part 3) - Dose-Adjusters (N=5)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 3 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 5 | 1 | 0 | 6 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 2 | 6 | 1 | 2 | 4 | 0 | 3 | 2 | 0 | 2 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 0 | 4 | 5 | 4 | 7 | 0 | 3 | 2 | 1 | 2 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 7 | 3 | 2 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 6 | 5 | 4 | 4 | 0 | 2 | 2 | 1 | 3 | 0
Fatigue (General disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 4 | 4 | 4 | 0 | 0 | 0 | 3 | 2 | 3 | 0
Seasonal allergy (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Ear infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 3 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 5 | 1 | 3 | 3 | 1 | 4 | 3 | 0 | 2 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 15 | 8 | 12 | 11 | 2 | 9 | 5 | 10 | 6 | 0
Otitis media (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngitis streptococcal (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 1
Rhinitis (Infections and infestations) | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 3 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 4 | 2 | 3 | 5 | 0 | 3 | 4 | 3 | 3 | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 3 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 2 | 2 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Weight increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0
Increased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 2 | 16 | 6 | 7 | 8 | 0 | 4 | 3 | 2 | 5 | 0
Poor quality sleep (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Psychomotor hyperactivity (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aggression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 2 | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 2 | 4 | 1 | 0
Impulsive behaviour (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2
Irritability (Psychiatric disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mood swings (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nightmare (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Stereotypy (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gynaecomastia (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 5 | 3 | 1 | 2 | 0 | 5 | 0 | 1 | 4 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 5 | 3 | 0 | 6 | 1 | 2 | 2 | 3 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 7 | 2 | 3 | 4 | 0 | 3 | 1 | 2 | 4 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 5 | 2 | 3 | 0 | 1 | 3 | 1 | 3 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Middle insomnia (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
Study was terminated early, therefore, there was limited data collected in Open Label Extension part of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2018-12-19): https://cdn.clinicaltrials.gov/large-docs/31/NCT02901431/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-14): https://cdn.clinicaltrials.gov/large-docs/31/NCT02901431/SAP_001.pdf